CLINICAL TRIAL: NCT01821274
Title: A 21-Day, Randomized, Controlled Study to Evaluate the Irritation Potential of Diltiazem Hydrochloride 2% Cream in Healthy Subjects, Using a Cumulative Irritant Patch Test Design
Brief Title: A 21-Day Topical Safety Study of Diltiazem Hydrochloride Using a Cumulative Irritant Patch Test Design
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ventrus Biosciences, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: VEN307-DERM-002
Record Dates: First submitted 2013-03-26; First posted 2013-03-29 (Estimated); Last update posted 2013-08-21 (Estimated); Status verified 2013-07

CONDITIONS: Skin Irritation
MeSH Terms: interventions — Diltiazem; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- topical Diltiazem Hydrochloride 2% Cream (Experimental): 0.2 g applied topically under occlusive patch conditions to the infrascapular area of the back, once daily for 21 consecutive days over 3 weeks.
  Interventions: Drug: Diltiazem Hydrochloride 2% Cream
- Vehicle Cream (Placebo Comparator): 0.2 g applied topically under occlusive patch conditions to the infrascapular area of the back, once daily for 21 consecutive days over 3 weeks.
  Interventions: Drug: Vehicle Cream
- 0.2% sodium lauryl sulfate (SLS) (Active Comparator): 0.2 mL applied topically under occlusive patch conditions to the infrascapular area of the back once daily for 21 days over 3 weeks, will serve as a positive control.
  Interventions: Drug: 0.1% solution o sodium lauryl sulfate (SLS)
- 0.9% saline (Placebo Comparator): 0.2 mL, applied topically under occlusive patch conditions to the infrascapular area of the back once daily for 21 days over 3 weeks, will serve as a negative control.
  Interventions: Drug: Saline 0.9%

INTERVENTIONS:
Drug: Diltiazem Hydrochloride 2% Cream — 0.2 g applied topically to the infrascapular area of the back.
  Arms: topical Diltiazem Hydrochloride 2% Cream
Drug: Vehicle Cream — 0.2 g (contains no active pharmaceutical ingredient) applied topically to the infrascapular area of the back.
  Arms: Vehicle Cream
Drug: 0.1% solution o sodium lauryl sulfate (SLS) — 0.2 mL applied topically to the infrascapular area of the back will serve as a positive control.
  Arms: 0.2% sodium lauryl sulfate (SLS)
Drug: Saline 0.9% — 0.2 mL applied topically to the infrascapular area of the back will serve as a negative control.
  Arms: 0.9% saline

SUMMARY:
The purpose of the study is to determine whether Diltiazem Hydrochloride 2% Cream will cause irritation to skin on the back of healthy volunteers after repeated application over 21-days.

DETAILED DESCRIPTION:
The primary objective of this study will be to determine the potential of Diltiazem Hydrochloride 2% Cream to cause irritation after repeated topical application to the healthy skin of humans under controlled conditions.

In addition, safety will be assessed by evaluation of any adverse events (AEs) reported during the study.

ELIGIBILITY:
Inclusion Criteria:

* Are healthy males or females (to be confirmed by medical history)
* Are 18 years of age or older
* In the case of females of childbearing potential, are using an acceptable form of birth control (oral/implant/injectable/transdermal contraceptives, intrauterine device, condom with spermicide, diaphragm with spermicide, abstinence, partner's vasectomy). Abstinence or vasectomies are acceptable if the female subject agrees to implement one of the other acceptable methods of birth control if her lifestyle/partner changes
* If a female of childbearing potential, have a negative urine pregnancy test (UPT) at Screening, and are willing to submit to a pregnancy test at end of study (EOS)
* Are free of any systemic or dermatologic disorder, which, in the opinion of the investigator, will interfere with the study results or increase the risk of adverse events
* Are of any skin type or race, providing the skin pigmentation will allow discernment of erythema
* Complete a Medical Screening form as well as a Medical Personal History form
* Read, understand, and provide signed informed consent

Exclusion Criteria:

* Have sick sinus syndrome except in the presence of a functioning ventricular pacemaker (confirmed via medical history
* Have second-or third-degree AV block except in the presence of a functioning ventricular pacemaker (confirmed via medical history)
* Have hypotension (less than 90 mm Hg systolic, determined by performing vital signs)
* Have acute myocardial infarction and pulmonary congestion documented by x-ray (confirmed via medical history)
* Have any visible skin disease at the application site which, in the opinion of the investigative personnel, will interfere with the evaluation of the test site reaction
* Are not willing to refrain from using systemic/topical analgesics such as aspirin (81 mg daily aspirin will be allowed), Aleve, Motrin, Advil, or Nuprin for 72 hours prior to Day 1 and during the study (occasional use of acetaminophen will be permitted)
* Are using systemic/topical corticosteroids for 3 weeks prior to and during the study, or systemic/topical antihistamines for 72 hours prior to Day 1 and during the study
* Are using medication which, in the opinion of the investigative personnel, will interfere with the study results, including anti-inflammatory medications
* Are unwilling or unable to refrain from the use of sunscreens, cosmetics, creams, ointments, lotions, or similar products on the back during the study
* Have psoriasis and/or active atopic dermatitis/eczema
* Are females who are pregnant, plan to become pregnant during the study, or are breast-feeding a child
* Have a known sensitivity to constituents present in the material being evaluated
* Have damaged skin in or around the test sites, including sunburn, excessively deep tans, uneven skin tones, tattoos, scars, excessive hair, numerous freckles, or other disfigurations of the test site
* Have received treatment for any type of internal cancer within 5 years prior to study entry
* Have a history of, or are currently being treated for skin cancer
* Are currently participating in any clinical testing
* Have any known sensitivity to adhesives
* Have received any investigational treatment(s) within 4 weeks prior to study entry

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-03; Primary Completion 2013-07 (Actual); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Mean cumulative irritation score of Diltiazem Hydrochloride 2% Cream in healthy skin of humans. | 21 days
  The primary variable of interest is the mean cumulative irritation score. The mean cumulative irritation score for each subject, product and site will be calculated as the sum of the irritation scores divided by the number of readings. The total cumulative irritation score for each subject and product will also be calculated as the sum of irritation scores on each of 21 evaluation days. A normalized total score for each patch will be calculated by summing the total irritation scores for all subjects, dividing by the number of readings and multiplying by 210. These parameters will be tested pairwise for product differences using Fisher's protected least significant differences in the context of the analysis of variance (ANOVA), including effects of subject and product (ie, randomized complete blocks). All pairwise differences will be tested. No adjustment for multiple comparisons will be made.

CONTACTS AND LOCATIONS:
Locations (1):
- TKL Research, Paramus, New Jersey, United States